CLINICAL TRIAL: NCT04563156
Title: Follow-up and Rehabilitation of Survivors of Severe Covid-19 Infection
Brief Title: Follow-up and Rehabilitation of Survivors of Severe Coronavirus Disease 2019 (COVID-19) Infection
Acronym: SegCov
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 4047553
Record Dates: First submitted 2020-09-23; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: COVID19; LUNG FUNCTION; QUALITY OF LIFE; REHABILITATION; RISK FACTOR; FOLLOW-UP
MeSH Terms: conditions — COVID-19 | interventions — Respiratory Function Tests; Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe Covid-19 Survivors: Severe Covid-19 survivors previously admitted in the hospital
  Interventions: Diagnostic Test: Lung Function Test

INTERVENTIONS:
Diagnostic Test: Lung Function Test — Lung Function Test at 1, 4, 6 and 12 months after discharge. Computerized tomography scan at 6 months after discharge. Cardiopulmonary Exercise Testing at 6 months after discharge
  Other Names: Computerized tomography scan; Cardiopulmonary Exercise Testing

SUMMARY:
Infection with covid-19 is associated with respiratory failure, which when related to other etiologies can lead to reduced quality of life, physical, cognitive and mental dysfunction. There is no knowledge of the possible consequences of severe covid-19 infection.

Our objective is to describe these repercussions, identifying risk factors and assessing the impact of physical training.

At least 100 patients over 18 years of age who survive severe Covid-19 infection will be evaluated. Assessments after 1, 4, 6 and 12 months after hospital discharge. Quality of life, dyspnea, activity of daily living, muscle strength, mental and cognitive dysfunction will be evaluated, as well as pulmonary function test, cardiopulmonary stress test and chest tomography. Return to work, thromboembolic events and mortality up to 12 months will also be monitored.

Hospitalization data will be used to identify factors related to quality of life, fatigue and respiratory dysfunction. Predefined risk factors will be evaluated: age, sex, smoking, previous comorbidities index, previous clinical frailty, serum C-reactive protein and leukocyte / lymphocyte ratio in the first 24 hours of hospitalization, time between onset of symptoms and hospitalization, ICU and mechanical ventilation, time on mechanical ventilation, compliance corrected by the ideal weight at the start of mechanical ventilation, driving pressure, tidal volume corrected by the ideal weight and PEEP (positive end expiratory pressure) after 24 hours of intubation in controlled ventilation, tidal volume corrected by the ideal weight after 24 hours of spontaneous ventilation, inspiratory muscle training and pulmonary rehabilitation after hospital discharge.

DETAILED DESCRIPTION:
Prospective longitudinal study in which survivors of severe infection with the covid-19 virus (need for hospitalization with supplementation of more than 3l / min of oxygen or mechanical ventilation) will be evaluated after 1 month, 4 months, 6 months and 1 year after hospital discharge through distance or face-to-face assessment.

Patients will be included according to a convenience sample until 12/31/2020 with follow-up until 12/31/2021. The EQ-5D questionnaire will be collected to assess quality of life. For other secondary outcomes, the clinical frailty scale, daily life independence scale, MoCA cognition questionnaire, hospital anxiety and depression questionnaire (HADS), muscle strength measure by the MRC scale, dyspnea measure by the mMRC and BDI scale will be used -TDI, 1-minute sit-and-stand test, maximum inspiratory and expiratory pressure measurement. Return to work, occurrence of thromboembolic events, occurrence of falls, need for re-hospitalization and mortality up to 12 months after admission will also be evaluated.

After 6 months of discharge, lung volume measurement will be performed by pulmonary function test, aerobic capacity by cardiopulmonary exercise test and evaluation of anatomical pulmonary sequelae by chest tomography. Patients residing close to the hospital will be offered a physical training program carried out by the physiotherapy team with assessment of functional response indicators.

The data obtained in the follow-up will be crossed with data obtained by the Epicov study in order to identify risk factors related to dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Respiratory infection confirmed by reverse-transcriptase polymerase chain reaction (RT-PCR) for SARS CoV-2 swab
* Need for admission to the ICU or ward with need for oxygen greater than 3L / min or mechanical ventilation and has been discharged from hospital.

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age whom was admitted at the Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (University of São Paulo Faculty of Medicine Clinics Hospital) with positive RT-PCR for SARS CoV-2 swab that needed oxygen supplementation greater than 3L / min or mechanical ventilation and has been discharged from hospital after improvement.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessment of a survivor of severe COVID-19 infection 6 months after hospital discharge; | 6 months after discharge
  EQ-5D is a standardized tool for the assessment of quality of life in 5 different dimensions (Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression). Possible scores range from 1 (No problem) to 3 (Extreme problems) and each dimension are evaluated individually. Assessment at 6 months after discharge

SECONDARY OUTCOMES:
Quality of life questionnaire EQ-5D | 30, 120 days and 12 months after hospital discharge
Evaluation of dyspnea by the Modified Medical Research Council Scale (mMRC) | 30, 120 days, 6 months and 12 months after hospital discharge
The Hospital Anxiety and Depression Scale | 6 months and 12 months after hospital discharge
Baseline and Transition Dyspnea Indexes (BDI-TDI) | 30 days, 120 days, 6 and 12 months after hospital discharge;
Clinical frailty scale measured after discharge from the ICU, | 30, 120 days, 6 and 12 months after hospital discharge
Lawton-Brody Instrumental Activities of Daily Living (iADL) scale | 30, 120 days, 6 months and 12 months after hospital discharge
Muscle strength according to the Medical Research Council (MRC) scale | 30, 120 days, 6 and 12 months after hospital discharge;
Maximum inspiratory pressure, diaphragmatic mobility and diaphragm thickness | 30, 120 days, 6 and 12 months after hospital discharge
Sit-to-stand test in 1 minute | 30 days, 120 days, 6 and 12 months after hospital
Cognitive dysfunction measured using the Montreal Cognitive Assessment (MoCA) test | 6 months and 12 months after hospital discharge
Pulmonary function test with Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) measurements | 30, 120 days and 6 and 12 months after hospital discharge
Hemoglobin, hematocrit, creatinine and Fasting plasma glucose (FPG) | 6 and 12 months after hospital discharge;
Quantitative computerized tomography scan | 6 months after hospital discharge
Maximum VO2 during Cardiopulmonary exercise testing | 6 and 12 months after hospital discharge
Return to work | 6 months and 12 months after hospital discharge
Occurrence of thromboembolic events after | 6 and 12 months after hospital discharge
Occurrence of falls | 6 and 12 months after hospital discharge
Need for readmission | 6 and 12 months after hospital discharge
Mortality | 6 and 12 months after hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo-HCFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toufen C Jr, Costa EL, Hirota AS, Li HY, Amato MB, Carvalho CR. Follow-up after acute respiratory distress syndrome caused by influenza a (H1N1) virus infection. Clinics (Sao Paulo). 2011;66(6):933-7. doi: 10.1590/s1807-59322011000600002. PMID 21808854
- [Background] Toufen Junior C, De Santis Santiago RR, Hirota AS, Carvalho ARS, Gomes S, Amato MBP, Carvalho CRR. Driving pressure and long-term outcomes in moderate/severe acute respiratory distress syndrome. Ann Intensive Care. 2018 Dec 7;8(1):119. doi: 10.1186/s13613-018-0469-4. PMID 30535520